CLINICAL TRIAL: NCT05515757
Title: Development of a Hospital-Based Contingency Management Intervention
Brief Title: Hospital-Based Contingency Management
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: CareOregon (Unknown); Affect Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Linda Peng, Principal Investigator, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00023484
Record Dates: First submitted 2022-08-10; First posted 2022-08-25 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Amphetamine-Related Disorders
Keywords: Amphetamine-Related Disorders; substance-related disorders; behavior therapy; psychology reinforcement; hospital medicine
MeSH Terms: conditions — Amphetamine-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile app-based contingency management (Other): All participants will be enrolled into an 8-week mobile app-based contingency management intervention starting during a prolonged hospitalization.
  Interventions: Behavioral: Mobile-app based contingency management

INTERVENTIONS:
Behavioral: Mobile-app based contingency management — We are adapting an evidence-based outpatient mobile-app based CM intervention to the hospital setting for hospitalized patients with stimulant use disorders requiring prolonged hospitalization. Participants will be enrolled into an 8-week mobile-app based contingency management intervention.

SUMMARY:
This study aims to adapt an outpatient mobile app-based contingency management intervention to the hospital setting to understand how we can use contingency management to improve health outcomes in hospitalized patients with stimulant use disorders.

DETAILED DESCRIPTION:
Contingency management (CM), an evidence-based strategy that utilizes a reward-based system as positive reinforcement, has been most robustly studied in the outpatient setting, but also has the potential to improve hospital care for patients with stimulant use disorder. The hospital is a challenging environment for people who use drugs. Conflicts with staff often result from in-hospital substance use, prolonged time off the unit, and missing medications, leading to negative health outcomes and re-admissions. By relying on positive rewards to encourage positive health behaviors, CM has the potential to improve staff-patient relationships, healthcare engagement, and reduce substance use in the hospital. Stimulant use disorder is especially difficult to address in the hospital due to a lack of medications that can support cravings and withdrawal symptoms. However, little is known about CM implementation in hospitals and the hospital setting may introduce unique challenges.

The objective of this study is to adapt an outpatient mobile app-based CM intervention to the hospital setting to understand the feasibility and acceptability of a hospital-based CM intervention to improve health outcomes in hospitalized patients with substance use disorders. We'll achieve this objective through following specific aims: Aim 1: Identify adaptations needed to implement an evidence-based outpatient mobile-app based CM intervention to the hospital setting for hospitalized patients with substance use disorders. Aim 2: Determine the feasibility, including facilitators and barriers, of implementing a mobile app-based CM intervention in the hospital setting. Aim 3: Assess the acceptability of a mobile app-based hospital-based CM intervention to patients and staff.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older
* Have moderate to severe stimulant use disorder, as diagnosed using DSM-5 criteria for stimulant use disorder by an addiction medicine provider
* Have an anticipated hospital length of stay greater than 2 weeks
* Be able to use a smartphone and agree to download and use the Affect app as part of study-related procedures
* Be English speaking and be able to understand explanations of study procedures and the informed consent to participate

Exclusion Criteria:

* Unable to engage in the intervention due to cognitive impairment or altered mental status
* Unable to engage in the intervention due to acute medical/mental health issues, per judgement of the research assistant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Intervention acceptability and feasibility | Week 0-8
  Evaluated using semi-structured qualitative interviews with participants and staff

SECONDARY OUTCOMES:
Brief Addiction Monitor (BAM) | Week 0-8
  The Brief Addiction Monitor (BAM) is a 17-item, multidimensional, progress-monitoring instrument for patients with a substance use disorder. The BAM includes items that assess risk factors for substance use, protective factors that support recovery, and drug and alcohol use. This instrument will be used to monitor the progress of the participants substance use disorder. Each functional domain of the survey (use, risk, protective) has an associated composite score which serves as a marker of clinical status. For Use (Scores 0 to 12), higher scores mean more substance use. For Risk (scores 0 to 24), higher sores mean more risk. For Protective (scores 0 to 24), higher scores mean more protection.
Participant engagement in the contingency management intervention | Week 0-8
  Participation in the contingency management intervention will be tracked. This includes number of counseling appointments attended and number of self-reflection activities attended. This is an implementation outcome where we measure how often participants are engaging in this intervention.
Participant drug test results | Week 0-8
  Participants can complete twice weekly drug testing as part of the contingency management intervention. We will measure the number of positive and negative drug tests as an objective measure of substance use.

CONTACTS AND LOCATIONS:
Locations (1):
- Linda Peng, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peng L, Young K, Titus H, Peeples J, Song E, DeFrancesco C, Roellich P, Phillips R, Englander H. Supporting Patients With Stimulant Use Disorder During and After Hospitalization With a Mobile App-based Contingency Management Intervention: A Feasibility and Acceptability Study. J Addict Med. 2025 Nov 25. doi: 10.1097/ADM.0000000000001621. Online ahead of print. PMID 41287143